CLINICAL TRIAL: NCT07039084
Title: A Randomized Cross-over Trial Examining the Efficacy of Implementing a Speech-generating Device for Childhood Dementia
Brief Title: Using a Speech-Generating Device to Support Communication in Childhood Dementia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 115839
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: Childhood Dementia; Genetic Disease; Nonverbal Communication; Augmentative and Alternative Communication
MeSH Terms: conditions — Genetic Diseases, Inborn; Nonverbal Communication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: As well as the outcome assessments, research assistants completing coding/rating and integrity/reliability assessments will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment then Control (Other): The arm receives the intervention (device), then the control
  Interventions: Device: Speech-generating device; Other: Control
- Control then Treatment (Other): The arm receives the control, then the treatment (device)
  Interventions: Device: Speech-generating device; Other: Control

INTERVENTIONS:
Device: Speech-generating device — The device is an iPad loaded with a grid-based and speech-generating communication application - a suitable application for the participant is determined at the beginning of the trial. This device is used in all 12 therapy sessions and implemented by a qualified speech pathologist in a natural, play-based setting.
  Other Names: augmentative and alternative communication; communication device
Other: Control — Participants will continue their current model of care. This means that if participants are receiving speech therapy locally, they may continue to do so given that no speech-generating device is introduced or used during this time. Participants will check in with the researching clinician at least once a week via telehealth or phone call - the aim is to stay in contact with families and reduce loss to follow-up. The clinician will also monitor treatment integrity and document any differences that may be present during this phase.
  Other Names: Usual care

SUMMARY:
Individuals with childhood dementia experience loss of developmental skills and many have limited verbal speech. The aim of this clinical trial is to examine how well a speech-generating device supports the communication skills of participants with childhood dementia. The speech-generating device is a communication program loaded onto an iPad.

This is a crossover trial, meaning that each participant will receive both the treatment (device) and a control (usual care; no device) phase. The order in which each participant receives the device versus the usual care (no device) will depend on which group the participant is assigned to. The changes in communication in each phase will then be compared.

During the trial, participants can expect to complete a series of assessments and attend a total of 2 x 1-hour therapy session per week for 6 weeks.

DETAILED DESCRIPTION:
The umbrella term 'childhood dementia' describes the hundreds of rare neurodegenerative genetic disorders occurring in children. Individuals with childhood dementia experience loss of developmental skills - many children have limited verbal speech to begin with but continue to lose their ability to communicate as the disease progresses. Augmentative and alternative communication (AAC) is one of the ways to support children with little speech and children with childhood dementia should have access to such tools as early as possible. However, the efficacy of high-tech AAC methods, such as speech generating devices, for children with childhood dementia has not been rigorously examined.

In this randomised cross-over trial, 38 participants with childhood dementia will be randomised into two groups (n=19 per group), which will determine the sequence of treatment delivery. The primary aim of this trial is to evaluate the efficacy of implementing a speech-generating device for communication in childhood dementia compared with their usual care (i.e. no device). Change in communication will be measured using a patient-defined outcome - this outcome is a 'communicative act' chosen at the beginning of the trial with participants and their family. This means that each participant will have an individualised communication outcome which will be targeted during treatment sessions and measured in assessment sessions. The secondary aims include parent-reported communication, family impact and language/communication competence.

Each participant will complete screening, preference testing and baseline assessments about 2-4 weeks before randomisation. Further assessments will be completed before and after each phase. For each participant, the change in assessment scores between the start and the end of each period will be calculated. The mean difference in the change in total score between the two periods will then be calculated.

Each participant is expected to be involved in the study for 12 weeks after randomisation. This is split into two phases (6 weeks each). In the treatment (device) phase, each participant will receive two 1-hour therapy sessions per week, for 6 weeks, with a communication device (or 12 x 1-hour therapy within a 6-week treatment phase). The device is implemented by a qualified speech pathologist on the project team and can occur at Murdoch Children's Research Institute or at the participants' home.

The control (usual care) phase involves another 6 weeks, however, no therapy sessions are provided by the project team. Weekly phone-call or telehealth check-ins will be performed to ensure things are going smoothly.

ELIGIBILITY:
Inclusion Criteria:

* Is between the ages of 3 and 12 years, inclusive, at the time of enrolment
* Has a genetically confirmed Childhood Dementia (via genetic report from a qualified geneticist), meeting the definition outlined in Elvidge et al. (2023) or is a condition listed on https://www.childhooddementia.org/what-is-childhood-dementia/childhood-dementia-disorders
* Passes a visual-motor screening test, therefore being able to tap on an iPad spontaneously or by imitation and has adequate hearing
* Considered "minimally verbal" with less than 20 spontaneous words (or gestalts) at baseline assessments, confirmed with the LVIS.
* Is not currently using a speech-generating device with proficiency (i.e. using the device as a main mode of communication on a daily basis).
* Is English-speaking or consents to therapy being conducted in English (parents will need to be able to complete the parent-reported measures in English)

Exclusion Criteria:

* Has an additional or dual genetic variation (as this is likely to cause multiple complications and increase variability),
* Is extremely ill or has progressed into a later stage of their disease (i.e. child has clinically significant loss of vision, hearing, fine motor skills, or is unable to adequately attend sessions due to illness),
* This is to ensure treatment is beneficial, reduce harm and reduce attrition rates.
* Lives outside of the state of Victoria (making it difficult for in-person appointments)
* Inability or unwillingness of participant or legally acceptable representative to give written informed consent.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Changes in the frequency of target communicative act related to the patient-defined outcome determined at the beginning of the trial | Baseline, Week 0, Week 6 and Week 12
  Each participant will have specific communicative acts related to a patient-defined outcome determined at the beginning of the trial with each participant and their family. This means that each participant will have an individualised communication outcome which will be targeted during treatment sessions. The change in frequency of these specific communicative acts will be measured. The mean difference of each period (comparing the start to end of the phase) will be determined and compared between the 2 periods.

SECONDARY OUTCOMES:
Changes in overall communicative acts | Baseline, Week 0, Week 6 and Week 12
  Changes in overall communicative acts measured through the difference in total number of all communicative acts observed between the two periods. This will be measured by the overall number of communicative acts observed during an assessment session regardless of the relation to the patient-defined outcome. The change in the total score between the start and the end of each period will be calculated for each participant. The mean difference in the change in total score between the two periods will then be calculated.
Changes in parent-reported communication via the Communication Matrix total score | Baseline, Week 0, Week 6 and Week 12
  Changes in parent-reported communication skills will be measured using the Communication Matrix total score. For each participant the change in the total score between the start and the end of each period will be calculated. The mean difference in the total score between the two periods will then be calculated. The Communication Matrix allows for the quantification of reported behaviours, e.g. the total score is calculated by scoring each cell in the Matrix (each cell representing a communication behaviour at a particular level of communication). Each cell is scored with 0 (Not used), 1 (Emerging - inconsistently used) or 2 (Mastered - used proficiently at all times). These points are summed to obtain a score between 0 to 160 and a percentage is obtained to represent the proportion of communication behaviours Mastered.
Changes in family and caregiver impact assessed via the Family Impact of Assistive Technology Scale for Augmentative and Alternative Communication (FIATS-AAC) | Baseline, Week 0, Week 6 and Week 12
  Changes in parent satisfaction, social impact and the mental health of caregivers will be assessed using the Family Impact of Assistive Technology Scale for Augmentative and Alternative Communication (FIATS-AAC). Each item is scored on a 7-point Likert scale and assigned into one of the 13 domains (Behavior, Caregiver Relief, Contentment, Doing Activities, Education, Energy, Face-to-Face Communication, Family Roles, Finances, Security, Self Reliance, Social Versatility, Supervision). The mean score for each domain (ranging between 1 to 7) are added together to produce the total score (ranging between 13 to 91). A higher domain score suggests a higher (more positive) functional level of that specific domain. The change in scores between the start and the end of each period will be calculated for each participant. The mean difference in the score between the two periods will then be calculated.
Changes in family and caregiver impact assessed via semi-structured interviews | Baseline, Week 6 and Week 12
  Changes in parent satisfaction, social impact and the mental health of caregivers will be assessed using a semi-structured interview as seen in Vogel et al. (2016), completed at baseline and at the end of each phase. Thematic analysis will be used to identify any themes that are present during these interviews and descriptively compare the differences identified.
Changes in Language / Communication Competence assessed via the Low-Verbal Investigatory Survey | Baseline, Week 0, Week 6 and Week 12
  Changes in the language and communication competence between the start and the end of each period for each participant will be determined via the Low-Verbal Investigatory Survey (LVIS). The survey produces a Verbal Communication score (between 0 to 15), an Alternative Communication score (between 0 to 11) and a Nonverbal Communication score (between 0 to 5). A higher score suggests greater communication competence in each of those areas. The mean differences in the LVIS scores between the two periods will then be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Murdoch Children's Research Institute, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data set collected for the analysis of this trial will be made available 12 months following analysis and publication of the primary outcome. The following will be made available long-term for use by future researchers from a recognised research institution:
  * Individual participant data that underlie the results reported after anonymisation/deidentification (text, tables, figures and appendices),
  * Trial protocol, Participant Information and Consent Form (PICF),
  * Statistical Analysis Plan (SAP), statistical code. Note that the data sharing of de-identified speech and language data is an Optional Consent for participants.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 12 months after publication of primary outcome
Access Criteria: Interested researchers may request access to the data by submitting a formal data sharing request to the Sponsor. The request will be reviewed by the Sponsor and the Sponsor-Investigator, and any relevant Murdoch Children's Research Institute (MCRI) data sharing committee, considering factors such as scientific merit, data security, and adherence to the approved research objectives. The data may be obtained from MCRI by emailing mctc@mcri.edu.au

REFERENCES:
- [Background] Ganz JB, Morin KL, Foster MJ, Vannest KJ, Genc Tosun D, Gregori EV, Gerow SL. High-technology augmentative and alternative communication for individuals with intellectual and developmental disabilities and complex communication needs: a meta-analysis. Augment Altern Commun. 2017 Dec;33(4):224-238. doi: 10.1080/07434618.2017.1373855. Epub 2017 Sep 19. PMID 28922953
- [Background] Nunn K, Williams K, Ouvrier R. The Australian Childhood Dementia Study. Eur Child Adolesc Psychiatry. 2002 Apr;11(2):63-70. doi: 10.1007/s007870200012. PMID 12033746
- [Background] Light J, McNaughton D. Communicative Competence for Individuals who require Augmentative and Alternative Communication: A New Definition for a New Era of Communication? Augment Altern Commun. 2014 Mar;30(1):1-18. doi: 10.3109/07434618.2014.885080. PMID 30952185
- [Background] Elvidge KL, Christodoulou J, Farrar MA, Tilden D, Maack M, Valeri M, Ellis M, Smith NJC; Childhood Dementia Working Group. The collective burden of childhood dementia: a scoping review. Brain. 2023 Nov 2;146(11):4446-4455. doi: 10.1093/brain/awad242. PMID 37471493
- See also: Conditions that cause childhood dementia — https://www.childhooddementia.org/what-is-childhood-dementia/childhood-dementia-disorders
- See also: Global research inequity and opportunities for childhood dementia — https://www.childhooddementia.org/news/report-reveals-global-research-inequity
- See also: Word Health Organisation: Global report on assistive technology — https://www.who.int/publications/i/item/9789240049451